CLINICAL TRIAL: NCT00116389
Title: An Open-Label Phase 2 Trial of Talabostat and Gemcitabine in Patients With Stage IV Adenocarcinoma of the Pancreas
Brief Title: Trial of Talabostat and Gemcitabine in Patients With Stage IV Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Hold May 2007
Sponsor: Point Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTH-320
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatic Cancer; Neoplasm Metastasis; Adenocarcinoma
Keywords: pancreatic cancer; cancer of the pancreas; adenocarcinoma of the pancreas; pancreatic neoplasms; Metastatic pancreatic cancer (Stage IV); Stage IV Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — PT-100 dipeptide; Gemcitabine

INTERVENTIONS:
Drug: talabostat mesylate tablets
Drug: gemcitabine

SUMMARY:
The purpose of this study is to assess the 6-month survival rate and safety of talabostat and gemcitabine in patients with stage IV adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥18 years
* Histologically confirmed metastatic (stage IV) adenocarcinoma of the pancreas
* Measurable disease defined per RECIST
* Karnofsky Performance Status ≥50
* Expected survival ≥12 weeks
* Provide written informed consent

Exclusion Criteria:

* CNS metastases
* Prior treatment with other chemotherapy for pancreatic cancer unless used as a radiosensitizer
* Radiation therapy to >25% of the bone marrow
* Clinically significant laboratory abnormalities
* Any malignancy within the 5 years immediately prior to the first dose of study medication with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix
* The need for chronic (i.e., >7 days) oral or intravenous corticosteroid therapy with >10mg/day prednisone equivalents
* Any comorbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol
* Patients who are within 28 days of radiation therapy, biologic therapy, immunotherapy, or other investigational medication. All side effects of prior treatment must have resolved at study entry.
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
6 month survival

SECONDARY OUTCOMES:
overall survival
progression-free survival (PFS)
quality of life
pain
performance status

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Northwest Alabama Cancer Center, PC, Florence, Alabama
  - Northwest Alabama Cancer Center, PC, Muscle Shoals, Alabama
  - Oncology Associates, PC, Hartford, Connecticut
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Cancer Center of Florida, Ocoee, Florida
  - Hematology Oncology Associates of Central Brevard, Rockledge, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Yagnesh V. Oza, MD, Mount Vernon, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - Cancer Care Center, Inc., New Albany, Indiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Huron Medical Center, Port Huron, Michigan
  - Billings Clinic, Billings, Montana
  - Monmouth Medical Center, Long Branch, New Jersey
  - New York Oncology Hematology/Albany Regional Cancer Center, Albany, New York
  - Hematology-Oncology Associates of Rockland, New City, New York
  - Dayton Oncology and Hematology, Kettering, Ohio
  - Lawrence M. Stallings, MD, Wooster, Ohio
  - Trilogy Cancer Center, Wooster, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Clinic, The, Portland, Oregon
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Oncology, PA, Presbyterian, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Elkins Pancreas Center, Houston, Texas
  - Saint Luke's Episcopal Hospital, Houston, Texas
  - Cancer Care Northwest, Spokane, Washington